CLINICAL TRIAL: NCT02558309
Title: Optic Nerve Head Quantification While Reducing Elevated Intracranial Pressure
Status: Withdrawn | Type: Observational
Why Stopped: The Primary Investigator is no longer with UPMC. No patients have been enrolled.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: PRO15070113
Record Dates: First submitted 2015-09-22; First posted 2015-09-23 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Intraocular Pressure; Intracranial Hypertension
MeSH Terms: conditions — Intracranial Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Intracranial Pressure Reduction: Subjects scheduled to undergo gradual, step-wise reduction of Intracranial Pressure (ICP) will be screened.
  * The Glasgow Coma Scale will be administered to ascertain the cognitive ability of the participant.
  * A slit lamp examination and indirect ophthalmoscopy will be performed.
  Experimental:
  * The subject's eye will be held open with an eye speculum during the exam.
  * Another eye exam, which includes a slit lamp examination and indirect ophthalmoscopy, will be performed.
  * Intraocular Pressure will be measured.
  * An Optic Coherence Tomography (OCT) will be performed.
  * At each step along the process of ICP reduction, the eye exam, IOP & OCT will be performed.
  Optional:
  * The Ophthalmology study team will raise the IOP using an Ophthlmodynanometer. It will be raised to 20 mmHg and 40 mmHg while OCT scans are obtained.
  * OCT scans will be taken at pre-manipulation, 20mmHg, 40mmHg, and post-manipulation at each step of the ICP lowering procedure.

SUMMARY:
The goal of this study is to examine in-vivo the effect of intraocular (IOP) and intracranial pressures (ICP) on the optic nerve head (ONH). The effect of ICP on eye health has been an area of concrete research effort in recent years. The ability to acquire non-invasive and highly detailed information on both the eye and the brain using technologies such as magnetic resonance imaging (MRI) and optical coherence tomography (OCT) have paved the way to assess non-invasively the effect of ICP in-vivo. In this study, we will quantify the structural changes in the ONH in subjects with elevated ICP while they are treated to reduce the elevated pressure. This process will occur in a stepwise fashion over a period of time determined by the clinical treatment plans. We will apply controlled pressures to the eye during each step of ICP lowering while OCT images are obtained.

DETAILED DESCRIPTION:
Objective:

The goal of this study is to examine in-vivo the effect of intraocular (IOP) and intracranial pressures (ICP) on the optic nerve head (ONH).

Specific Aims:

In this study, the investigators will quantify the structural changes in the ONH in subjects with elevated ICP while they are treated to reduce the elevated pressure. This process will occur in a stepwise fashion over a period of time determined by the clinical treatment plans. The investigators will apply controlled pressures to the eye during each step of ICP lowering while OCT images are obtained.

Background:

The effect of ICP on eye health has been an area of concrete research effort in recent years. The ability to acquire non-invasive and highly detailed information on both the eye and the brain using technologies such as magnetic resonance imaging (MRI) and optical coherence tomography (OCT) have paved the way to assess non-invasively the effect of ICP in-vivo.

The ONH separates two pressurized compartments: the eyeball and the central nervous system. Situations in which ICP is elevated are often associated with papilledema, though the magnitude and the rate of change in ONH elevation in response to increased ICP or the reduction in ONH elevation in response to ICP treatments are yet to be determined. On the opposite side, glaucoma is a leading cause of blindness where elevated IOP is the leading risk factor, with clinical evidence suggesting the presence of ICP below the normal level in these subjects. The impaired balance between IOP and ICP leads to the deformation of the ONH, which triggers strangulation of the retinal ganglion cell axons when trespassing through the lamina cribrosa within the ONH on their way from the eye to the brain, leading to gradual axonal loss and irreversible visual impairment.

Significance:

Little is known about how the interaction of IOP and ICP pressure changes affect the macrostructure and microstructure of the optic nerve head structure. This information has a significant impact both for neurosurgical conditions with elevated ICP along with ocular conditions such as glaucoma and papilledema. The ability to gauge non-invasively changes in ICP will have a tremendous impact on neurosurgical management as it eliminates the need of longitudinal invasive measurements of ICP. The study will also improve the investigator's understanding of the pathophysiologic processes that lead to development of glaucoma as well as the response to treatment for subjects with papilledema. A better understanding of these processes will ultimately lead to improved detection and management of these conditions and a better understanding of ocular bio-mechanics.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older.
* Patients with an external ventricular drain (EVD).
* Normally appearing eye as determined during the screening clinical examination.

Exclusion Criteria:

* History of intraocular surgery or ocular trauma (with the exception of laser procedures or uneventful cataract surgery more than 1 year from enrollment date).
* Ocular disorders that could affect retinal function such as retinal detachment, diabetic retinopathy, Macular degeneration.
* Neurological & Non-Glaucomatous causes for Visual Field damage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are scheduled to undergo gradual, step-wise reduction of Intracranial Pressure (ICP) will be screened.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-10; Primary Completion 2016-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Optic Nerve Head | 1 Week
  The optic nerve head (ONH) structures will be evaluated for tissue deformation. The association between the structural findings in the optic nerve head region and intracranial and intraocular pressures will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Gadi Wollstein, MD, Principal Investigator — University of Pittsburgh Medical Center